CLINICAL TRIAL: NCT03030040
Title: A Randomised Controlled Trial of a Mindfulness-based Cognitive Therapy Self-help Intervention for UK National Health Service Employees
Brief Title: A Randomised Controlled Trial of Self-help Mindfulness-based Cognitive Therapy for Health Workers
Acronym: MindSHINE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Sussex Partnership NHS Foundation Trust (Other); University of Sussex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EmilyIronmongerMRP2016; IRAS ID: 215054 (Other: UK National Health Service Health Research Authority)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Psychological Stress
Keywords: mindfulness-based cognitive therapy; self-help; healthcare staff
MeSH Terms: conditions — Stress, Psychological | interventions — Fumigant 93

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Random allocation of participants to arms will be conducted by a statistician independent of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT-SH (Experimental): MBCT-SH will be an unguided, mindfulness-based cognitive therapy, book-based self-help intervention.
  Interventions: Behavioral: The self-help book: Williams, M. & Penman, D. (2011). Mindfulness: A practical guide to finding peace in a frantic world. London: Piatkus.
- Control (No Intervention): A wait list control group who will receive no intervention during the 21 weeks of the study. Control participants will be provided with the self-help book that the MBCT-SH group received after week 21.

INTERVENTIONS:
Behavioral: The self-help book: Williams, M. & Penman, D. (2011). Mindfulness: A practical guide to finding peace in a frantic world. London: Piatkus. — Participants will be provided with a copy of the self-help book, and asked to read it and follow the activities outlined in it, over eight weeks. They will receive weekly standardized emails, to provide information about mindfulness and encouragement to engage with the self-help book.
  Arms: MBCT-SH

SUMMARY:
This study examines whether a mindfulness-based self-help book is effective at reducing healthcare workers' levels of stress and improving their wellbeing.

DETAILED DESCRIPTION:
This study is a randomised controlled trial (RCT) examining the efficacy of a mindfulness-based cognitive therapy self-help book ('Mindfulness: A practice guide to finding peace in a frantic world') relative to a wait-list control, in healthcare staff. It builds on a previous pilot RCT (http://www.isrctn.com/ISRCTN16486066). A battery of measures will be administered at baseline (week 0), post-intervention (week 9) and follow-up (week 21). This trial is designed to test the following hypotheses.

Primary Hypothesis

-Mindfulness-based cognitive therapy self-help (MBCT-SH) participants, in comparison to waitlist control participants, will show a reduction in symptoms of stress by the end of MBCT-SH (week 9).

Secondary Hypotheses

* The improvement detailed in the primary hypothesis will be maintained at a follow-up 12 weeks after the end of the MBCT-SH (week 21).
* MBCT-SH participants, in comparison to waitlist control participants, will show improvements in mindfulness, other-compassion, self-compassion, anxiety, depression, burnout and mental well-being by the end of MBCT-SH (week 9), and these improvements will be maintained at a follow-up 12 weeks after the end of the MBCT-SH (week 21).
* MBCT-SH participants, in comparison to waitlist control participants, will show a reduction in the number of sickness absence days from the three months preceding the intervention to the three months following the intervention.
* Increases in self-compassion and mindfulness from week 0 to week 9, will mediate the effects of MBCT-SH (relative to waitlist control) on levels of stress, depression, anxiety, wellbeing and burnout.

ELIGIBILITY:
Inclusion Criteria:

1. Being currently employed by Sussex Partnership NHS Foundation Trust (in the UK) in a role or roles that involve direct delivery of healthcare.
2. Having at least one day per week of direct contact with UK National Health Service service users.
3. Agreeing to refrain from engaging in another form of psychological therapy during the course of the study.
4. Having self-reported sufficient English language reading ability to read and understand the self-help book

Exclusion Criteria:

1. Being currently on leave of absence from work.
2. Having previously received a minimum dose (defined as 50% of a course or more) of a mindfulness-based intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Stress | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Stress sub-scale of the Depression, Anxiety and Stress Scale-21

SECONDARY OUTCOMES:
Stress (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Stress sub-scale of the Depression, Anxiety and Stress Scale-21
Depression | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Depression sub-scale of the Depression, Anxiety and Stress Scale-21
Depression (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Depression sub-scale of the Depression, Anxiety and Stress Scale-21
Anxiety | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Anxiety sub-scale of the Depression, Anxiety and Stress Scale-21
Anxiety (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Anxiety sub-scale of the Depression, Anxiety and Stress Scale-21
Compassion for others | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Compassion Scale
Compassion for others (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Compassion Scale
Self-compassion | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Self-compassion Scale - Short Form
Self-compassion (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Self-compassion Scale - Short Form
Mindfulness | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Five-Facet Mindfulness Questionnaire - Short Form
Mindfulness (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Five-Facet Mindfulness Questionnaire - Short Form
Burnout | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Maslach Burnout Inventory
Burnout (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Maslach Burnout Inventory
Mental Wellbeing | Post-intervention (i.e. 9-weeks after baseline)
  Change from baseline at 9-weeks on the Short Warwick-Edinburgh Mental Well-being Scale
Mental Wellbeing (follow-up) | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline at 21-weeks on the Short Warwick-Edinburgh Mental Well-being Scale
Sickness absence | Follow-up (i.e. 21 weeks after baseline)
  Change from baseline in the number of days of sickness absence over the previous 12 weeks at 21 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Emily C Ironmonger, MSc, Principal Investigator — Canterbury Christ Church University; Clara Strauss, PhD, Study Director — Sussex Partnership NHS Foundation Trust & University of Sussex; Kate Cavanagh, PhD, Study Director — University of Sussex; Fergal Jones, PhD, Study Director — Canterbury Christ Church University & Sussex Partnership NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Oxleas NHS Foundation Trust, Dartford, Kent
  - Sussex Partnership NHS Foundation Trust, Hove, Sussex

IPD SHARING:
Plan to Share IPD: No